CLINICAL TRIAL: NCT03588975
Title: A Prospective, Open-label, Randomized, Concurrent Active-controlled, Longitudinal, Multicenter, Phase 3 Clinical Study of the Safety and Efficacy of MACI in Patients Aged 10 to 17 Years With Symptomatic Chondral or Osteochondral Defects of the Knee
Brief Title: A Study of MACI in Patients Aged 10 to 17 Years With Symptomatic Chondral or Osteochondral Defects of the Knee
Acronym: PEAK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vericel Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 55-1702-1
Record Dates: First submitted 2018-04-04; First posted 2018-07-17 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chondral Defect; Osteochondritis Dissecans (OCD); Articular Cartilage Defect; Articular Cartilage Disorder of Knee
Keywords: OCD; cartilage; cartilage defect
MeSH Terms: conditions — Osteochondritis Dissecans | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MACI (Experimental): autologous cultured chondrocytes on porcine collagen membrane
  Interventions: Biological: MACI
- microfracture (Active Comparator): surgical procedure
  Interventions: Procedure: microfracture

INTERVENTIONS:
Biological: MACI — autologous cultured chondrocytes on porcine collagen membrane
  Arms: MACI
Procedure: microfracture — Arthroscopic microfracture treatment
  Arms: microfracture

SUMMARY:
The objective of this study is to compare the efficacy and safety of MACI® vs arthroscopic microfracture in the treatment of patients aged 10 to 17 years with symptomatic articular chondral or osteochondral defects of the knee.

DETAILED DESCRIPTION:
This is a 2-year prospective, multicenter, randomized, open-label, parallel group clinical trial; a total of 45 patients, ages 10 to 17 years, will be randomized to receive a 1-time treatment with MACI or microfracture (2:1, 30 MACI:15 microfracture).

After meeting screening criteria at the initial visit, all patients will have a screening arthroscopy to further assess study eligibility. During the screening arthroscopy, patients will be further evaluated against entry criteria. Cartilage lesion size will be measured prior to any cartilage repair procedure and randomization. All patients who meet the eligibility criteria and are considered suitable for treatment in the study will have a cartilage biopsy taken prior to randomization to study treatment. Eligible patients will be randomized during the screening arthroscopy procedure to receive either MACI or microfracture treatment. Patients randomized to microfracture will undergo the procedure during the screening arthroscopy.

All biopsied tissue will be sent to the Vericel manufacturing facility in Cambridge, Massachusetts, where the sample will be processed to isolate the autologous chondrocytes. Cells from patients randomized to the MACI group will be used in the preparation of the MACI implant; cells from patients randomized to the microfracture group will be cryopreserved.

Patients randomized to treatment with MACI will return within 12 weeks of the screening arthroscopy to undergo the chondrocyte implantation procedure via arthrotomy. Patients are to follow a recommended postoperative rehabilitation program and compliance with the rehabilitation schedule will be monitored.

Patients will be followed post-study treatment for 2 years (104 Weeks).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cartilage or osteochondral defects
* One or more International Cartilage Repair Society (ICRS) Grade III or IV chondral or unsalvageable osteochondral defects located on the femoral condyles and/or trochlea amenable to treatment with the surgical procedure determined at randomization (MACI or microfracture).
* At least 1 defect size ≥1.5 cm2 on the femoral condyles and/or the trochlea; defects include OCD lesions with a bone lesion depth of ≤6 mm and does not require a bone graft.
* Stable target knee (i.e., anterior and posterior cruciate ligaments should be free of laxity as well as stable and intact). Ligament repair or reconstruction procedures are allowed prior to screening arthroscopy.
* Intact meniscus or partial meniscus (at least 50% of functional meniscus remaining) in the target knee.

Exclusion Criteria:

* Any surgery on the target knee joint within 6 months prior to Screening (not including diagnostic arthroscopy)
* ICRS Grade III or IV chondral or unsalvageable osteochondral defects located on the patella or tibia or any lesion that is bipolar to the index lesion
* Concomitant inflammatory disease or other conditions that affects the joints (eg, rheumatoid arthritis, metabolic bone disease, psoriasis, symptomatic chondrocalcinosis)
* Known history of septic arthritis in the index knee joint
* Known history of hypersensitivity to gentamicin, other aminoglycosides, or products of porcine or bovine origin
* Females who are pregnant or lactating

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Who Achieve at Least a 10-point Improvement From Baseline in KOOS-Child Pain and Function (Sports and Recreational Activities) Scores | Baseline and Week 104
  A responder is defined as a participant with at least a 10-point change (improvement) in both the KOOS-Child Pain and Function (Sports and Recreational activities) scores from Baseline scores. The Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL).

SECONDARY OUTCOMES:
Change from Baseline in KOOS-Child subscores | Baseline and Week 104
  The Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL).
Change from Baseline in KOOS-Child subscores | Baseline and Week 52
  The Knee and Osteoarthritis Outcome Score for Children (KOOS-Child) is a validated knee-specific instrument developed to assess the patients' opinion of their knee and associated problems. KOOS consists of 5 subscales: Pain, Function in sports and recreational activities, other Symptoms, Function in activities of daily living (ADL), and knee related Quality of life (QOL).

OTHER OUTCOMES:
Treatment Emergent Adverse Events | Week 104
  A treatment emergent untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hopper, Study Director — Vericel Corporation
Locations (12):
- United States (12):
  - Stanford University, Palo Alto, California
  - Shriner's Hospital for Children Northern California, Sacramento, California
  - University of California Davis Health, Sacramento, California
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Akron Children's Hospital, Akron, Ohio
  - The Ohio State University Jameson Crane Sports Medicine Institute, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Penn Sports Medicine Center, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vericel Clinical Trial for Cartilage Repair — https://www.vcel.com/clinical-development/